CLINICAL TRIAL: NCT05207371
Title: Phase I / II Clinical Trial of GAIA-102 for Advanced and Relapse NSCLC
Brief Title: Clinical Trial of GAIA-102 for Advanced and Relapse NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GAIA BioMedicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAIA-102-LC01
Record Dates: First submitted 2021-11-19; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cell Therapy; NSCLC
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAIA-102 alone (Experimental): GAIA-102: 1 vial (2 x 10^8 cells) / dose at a fixed dose, 1 to 3 doses / week for 3 consecutive weeks.
  Interventions: Biological: Biological
- GAIA-102 with Pembrolizumab (Experimental): GAIA-102: 1 vial (2 x 10^8 cells) / dose at a fixed dose, 1 to 3 doses / week for 3 consecutive weeks.
  Pembrolizumab：200 mg Administer on Day 1.
  Interventions: Biological: Biological

INTERVENTIONS:
Biological: Biological — Intravenous injection of GAIA-102 alone or with Pembrolizumab (KEYTRUDA®︎)

SUMMARY:
Phase I Part :

Confirm the safety of GAIA-102 alone or GAIA-102 with pembrolizumab for advanced / relapse non-small cell lung cancer, and decide recommended dose for Phase II.

Phase II Part :

Explore the efficacy and safety of GAIA-102 alone or GAIA-102 with pembrolizumab for advanced / relapse non-small cell lung cancer at the recommended dose of GAIA-102 decided in the Phase I part.

DETAILED DESCRIPTION:
Phase I Part :

The GAIA-102 cohort (Level A1~A3) and the GAIA-102 + Pembrolizumab cohort (Level B1~B3) will be implemented in a 3 + 3 design. First, start from Level A1 and set the DLT evaluation period until Day 28 of Cycle 1, and confirm the safety up to Cycle 1_Day 28 of Level A1. After that, Level A2 and Level B1 will be started in parallel. After that, unless MTD is recognized, the safety at each level will be confirmed in sequence, and the recommended doses of Phase II part will be determined.

Phase II Part :

At the recommended number of doses confirmed in Phase I Part, 20 patients will be administered up to 3 cycles, and the safety and efficacy of GAIA-102 alone or with pembrolizumab will be evaluated by ORR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been confirmed to have NSCLC by histological or cytological examination
2. Patients with ECOG performance status (PS) 0-1 at the time of obtaining consent
3. Patients aged 20 years or older at the time of obtaining consent

Exclusion Criteria:

1. Patients with symptomatological cranial nerve system metastasis. If treatment for cranial nerve system metastasis has already been performed and the neurologically recovered state has been maintained for 2 weeks or more before registration, registration is possible.
2. Patients diagnosed with cancerous meningitis
3. Patients who received allogeneic hematopoietic stem cell transplantation
4. Patients with active autoimmune disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase I part | Cycle 1 (Cycle period is 28 days)
  Dose Limiting Toxicity
Phase II part | Week 26
  Objective Response Rate (%)

SECONDARY OUTCOMES:
Phase I part | Week 26
  * Objective Response Rate
  * Disease Control Rate
Phase I part | 2 year
  * Progression-free Survival
  * Overall Survival
Phase II part | 2 year
  * Progression-free Survival
  * Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Yoshikazu Yonemitsu, MD, PhD, Study Director — Graduate School of Pharmaceutical Sciences, Kyushu University
Locations (3):
- Japan (3):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka